CLINICAL TRIAL: NCT06128070
Title: Phase 2a Study of Adding Ruxolitinib With Tacrolimus/Methotrexate Regimen for Graft-versus-Host Disease Prophylaxis in Myeloablative Conditioning Hematopoietic Cell Transplantation in Pediatric and Young Adult Patients
Brief Title: Ruxolitinib With Tacrolimus and Methotrexate for the Prevention of Graft Versus Host Disease in Pediatric and Young Adult Patients Undergoing Allogeneic Hematopoietic Cell Transplant for Acute Myeloid Leukemia, Acute Lymphoblastic Leukemia, or Myelodysplastic Syndrome
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: City of Hope Medical Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 23010; NCI-2023-07401 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 23010 (Other: City of Hope Medical Center); P30CA033572 (NIH)
Record Dates: First submitted 2023-10-27; First posted 2023-11-13 (Actual); Last update posted 2025-10-31 (Actual); Status verified 2025-10

CONDITIONS: Acute Lymphoblastic Leukemia; Acute Myeloid Leukemia; Myelodysplastic Syndrome
MeSH Terms: conditions — Precursor Cell Lymphoblastic Leukemia-Lymphoma; Leukemia, Myeloid, Acute; Myelodysplastic Syndromes | interventions — Specimen Handling; Stem Cell Transplantation; Hematopoietic Stem Cell Transplantation; Methotrexate; merphos; ruxolitinib; Tacrolimus

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Prevention (Ruxolitinib, tacrolimus, methotrexate) (Experimental): Patients receive ruxolitinib PO BID from day -1 to day +100, tacrolimus IV on day -1, and methotrexate IV on days +1, +3, +6, and +11, and undergo HCT on day 0. Patients also undergo chest CT and ECHO/MUGA at screening and undergo collection of blood samples throughout the trial.
  Interventions: Procedure: Biospecimen Collection; Procedure: Chest Computed Tomography; Procedure: Echocardiography; Procedure: Hematopoietic Cell Transplantation; Drug: Methotrexate; Procedure: Multigated Acquisition Scan; Drug: Ruxolitinib Phosphate; Drug: Tacrolimus

INTERVENTIONS:
Procedure: Biospecimen Collection — Undergo blood sample collection
  Other Names: Biological Sample Collection; Biospecimen Collected; Specimen Collection
Procedure: Chest Computed Tomography — Undergo chest CT
  Other Names: Chest CT; Computed Tomography of the Chest
Procedure: Echocardiography — Undergo ECHO
  Other Names: EC
Procedure: Hematopoietic Cell Transplantation — Undergo HCT
  Other Names: HCT; Hematopoietic Stem Cell Infusion; Hematopoietic Stem Cell Transplantation; HSCT; SCT; Stem Cell Transplant; stem cell transplantation; Stem Cell Transplantation, NOS
Drug: Methotrexate — Given IV
  Other Names: Abitrexate; Alpha-Methopterin; Amethopterin; Brimexate; CL 14377; CL-14377; Emtexate; Emthexat; Emthexate; Farmitrexat; Fauldexato; Folex; Folex PFS; Lantarel; Ledertrexate; Lumexon; Maxtrex; Medsatrexate; Metex; Methoblastin; Methotrexate LPF; Methotrexate Methylaminopterin; Methotrexatum; Metotrexato; Metrotex; Mexate; Mexate-AQ; MTX; Novatrex; Rheumatrex; Texate; Tremetex; Trexeron; Trixilem; WR-19039
Procedure: Multigated Acquisition Scan — Undergo MUGA
  Other Names: Blood Pool Scan; Equilibrium Radionuclide Angiography; Gated Blood Pool Imaging; Gated Heart Pool Scan; MUGA; MUGA Scan; Multi-Gated Acquisition Scan; Radionuclide Ventriculogram Scan; Radionuclide Ventriculography; RNVG; SYMA Scanning; Synchronized Multigated Acquisition Scanning
Drug: Ruxolitinib Phosphate — Given PO
  Other Names: INCB-18424 Phosphate; Jakafi; Jakavi
Drug: Tacrolimus — Given IV
  Other Names: FK 506; FK-506; Fujimycin; Hecoria; Prograf; Protopic; Tacforius

SUMMARY:
This phase II trial tests how well ruxolitinib with tacrolimus and methotrexate work to prevent the development of graft versus host disease in pediatric and young adult patients undergoing allogeneic hematopoietic cell transplant for acute myeloid leukemia, acute lymphoblastic leukemia, or myelodysplastic syndrome. Ruxolitinib is a type of medication called a kinase inhibitor. It works by blocking the signals of cells that cause inflammation and cell proliferation, which may help prevent graft versus host disease (GVHD). Tacrolimus is a drug used to help reduce the risk of rejection by the body of organ and bone marrow transplants by suppressing the immune system. Methotrexate stops cells from making DNA, may kill cancer cells, and also suppress the immune system, which may reduce the risk of GVHD. Giving ruxolitinib with tacrolimus and methotrexate may prevent GVHD in pediatric and young adults undergoing allogeneic hematopoietic cell transplants.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Determine if the addition of ruxolitinib phosphate (ruxolitinib) to tacrolimus and methotrexate as graft-versus-host disease (GVHD) prophylaxis, is safe in pediatric and young adult patients with hematologic malignancies who are eligible to undergo allogeneic hematopoietic cell transplantation (HCT) from a matched donor. (Safety lead-in segment) II. Following a patient safety lead-in, evaluate the efficacy of ruxolitinib, when given as part of reduced intensity HCT from a matched related/unrelated donor, as assessed by 1 year graft-versus-host disease-free and relapse-free (GRFS) rates in pediatric and young adult patients. (Phase II segment)

SECONDARY OBJECTIVES:

I. Estimate the cumulative incidence of acute GVHD (aGVHD) and non-relapse mortality (NRM) at 100-days after transplant.

II. Estimate the cumulative incidence of chronic GVHD (cGVHD) at 1- and 2-years after transplant.

III. Estimate the probabilities of overall and progression-free survival (OS/PFS) at 1- and 2-years after transplant.

IV. Estimate the relapse/progression rate. V. Estimate rate of infection and development of second malignancies including lymphoproliferative disorders at 1- and 2-years post-transplant.

VI. Further evaluate the safety of this regimen by assessing:

VIa. Adverse event type, frequency, severity, attribution, time-course, and duration; VIb. Complications including: infection, and delayed engraftment.

EXPLORATORY OBJECTIVES:

I. Characterize and evaluate hematologic recovery, donor cell engraftment and immune reconstitution by cell count and flow cytometry of lymphocyte subsets.

II. Characterize changes in aGVHD biomarkers (Reg-3alpha, sTNF RI, IL2Ralpha), JAK-regulated pro-inflammatory cytokines (i.e. IL-6, TNFalpha, C-reactive protein [CRP], beta2Microglubuolin) and STAT3 phosphorylation (downstream of JAK signaling) over time and by aGVHD status/grade.

III. Evaluate the pharmacokinetics of ruxolitinib in pediatric and young adult patients.

OUTLINE:

Patients receive ruxolitinib orally (PO) twice daily (BID) from day -1 to day +100, tacrolimus intravenously (IV) on day -1, and methotrexate IV on days +1, +3, +6, and +11, and undergo HCT on day 0. Patients also undergo chest computed tomography (CT) and echocardiography (ECHO)/multigated acquisition scan (MUGA) at screening and undergo collection of blood samples throughout the trial.

After completion of study treatment, patients are followed up at 30 days after the last dose of ruxolitinib and at 1 and 2 years post transplant.

ELIGIBILITY:
Inclusion Criteria:

* Documented informed consent of the participant and/or legally authorized representative

  * Assent, when appropriate, will be obtained per institutional guidelines
* Agreement to allow the use of archival tissue from diagnostic tumor biopsies

  * If unavailable, exceptions may be granted with study primary investigator (PI) approval
* Age: 2-22
* Weight ≥25kg
* Eastern Cooperative Oncology Group (ECOG) ≤ 2
* Performance status: Karnofsky ≥ 60% for patients ≥ 16 years old OR Lansky status ≥ 60% for patients < 16 years old
* Candidate for allogeneic bone marrow transplant with and available matched related donor (MRD) or an 8/8 matched unrelated donor (MUD) who is willing to donate bone marrow (BM) or mobilized peripheral blood stem cells

  * Note: Donor selection process will be in accordance with City of Hope (COH)-standard operating procedures (SOPs) (B.001.09 Allogeneic Cellular Therapy Product Donor Evaluation, Selection & Consent), which follows Food and Drug Administration (FDA) guidelines for donation of hematopoietic stem/progenitor cells (HPCs) obtained from peripheral blood or bone marrow
* Diagnosis of acute leukemia (acute myeloid leukemia [AML] or acute lymphoblastic leukemia [ALL]) in complete remission, or myelodysplastic syndrome (MDS)
* Fully recovered from the acute toxic effects (except alopecia) to ≤ grade 1 from prior anti-cancer therapy
* Women of childbearing potential (WOCBP): negative urine or serum pregnancy test. If the urine test is positive or cannot be confirmed as negative, a serum pregnancy test will be required (to be performed within 30 days prior to day 1 of protocol therapy)
* Agreement by females and males of childbearing potential to use an effective method of birth control or abstain from heterosexual activity for the course of the study through at least 6 months after the last dose of protocol therapy

  * Childbearing potential defined as not being surgically sterilized (men and women) or have not been free from menses for > 1 year (women only)

Exclusion Criteria:

* Autologous stem cell transplant within 1 year prior to day 1 of protocol therapy
* Prior allogeneic transplantation
* Chemotherapy, radiation therapy, biological therapy, immunotherapy within 14 days prior to day 1 of protocol therapy

  * Note: Conditioning regimen within 21 days prior to day 1 of protocol therapy is not considered as an exclusion criterion.
  * Note: Patients on maintenance chemotherapy with agents listed are not excluded
* Herbal medications
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to study agent
* History of active tuberculosis
* Patients with history of thrombosis including but not limited to myocardial infarction (MI)/stroke and pulmonary embolism (PE)/deep vein thrombosis (DVT) within 6 months of enrollment
* Active diarrhea due to inflammatory bowel disease or malabsorption syndrome
* Clinically significant uncontrolled illness
* Active, uncontrolled systemic infection (viral, bacterial, or fungal) requiring antibiotics
* Known history of immunodeficiency virus (HIV) or hepatitis B or hepatitis C infection
* Other active malignancy
* Females only: Pregnant or breastfeeding
* Any other condition that would, in the investigator's judgment, contraindicate the patient's participation in the clinical study due to safety concerns with clinical study procedures
* Prospective participants who, in the opinion of the investigator, may not be able to comply with all study procedures (including compliance issues related to feasibility/logistics)

Ages: 2 Years to 22 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 40 (Estimated)
Dates: Start 2024-07-16 (Actual); Primary Completion 2030-11-22 (Estimated); Study Completion 2030-11-22 (Estimated)

PRIMARY OUTCOMES:
Incidence of adverse events | Up to day +30 post hematopoietic cell transplant (HCT)
  Defined using the modified Bearman Scale and the National Cancer Institute Common Terminology Criteria for Adverse Events version 5.0 scale.
Graft-versus-host disease (GVHD)-free and relapse-free (GRFS) | From the date of transplantation to the first time of observing the following events: grade 3-4 acute GVHD, chronic GVHD requiring systemic treatment, relapse, or death, assessed at 1 year post transplantation
  Will be estimated using the product-limit method of Kaplan and Meier.

SECONDARY OUTCOMES:
Patients receiving planned doses of ruxolitinib (feasibility) | At completion of therapy (up to day+100)
  Patients who have received at least 80% of planned doses of ruxolitinib are deemed to meet feasibility criteria.
Incidence of acute GVHD | At 100 days post HCT transplant
  Will be graded and staged according to Mount Sinai Acute GVHD International Consortium criteria. Will be estimated using the method described by Gooley et al (1999).
Incidence of non-relapse mortality | At 100 days post HCT transplant
  Defined as death occurring in a patient from causes other than relapse or progression. Will be estimated using the method described by Gooley et al (1999).
Incidence of chronic GVHD | At 1 and 2 years post HCT transplant
  Will be evaluated and scored according to National Institutes of Health Consensus Staging. Will be estimated using the method described by Gooley et al (1999).
Overall survival | From the day of stem cell infusion until death, up to 2 years
  Will be estimated using the product-limit method of Kaplan and Meier.
Progression free survival | From the date of stem cell infusion to the date of death, disease relapse/progression, whichever occurs first, up to 2 years
  Will be estimated using the product-limit method of Kaplan and Meier.
incidence of relapse/progression | From day of stem cell infusion (day 0) to first observation of disease relapse/progression, up to 2 years
  Will be estimated using the method described by Gooley et al (1999).
Infection rate | From day -1 to day 130 post HCT transplant
  Will be reported by site of disease, date of onset, severity and resolution, if any.
Incidence of secondary malignancies | From day of stem cell infusion (day 0) to first observation of event of interest, assessed at 1 and 2 years post HCT transplant
Hematologic recovery, donor cell engraftment and immune reconstitution | Up to 2 years
  Assessed using: absolute neutrophil count ≥ 0.5 x 10^3/uL achieved and sustained for 3 consecutive lab values on different days with no subsequent decline; platelets ≥ 20 K/uL independent of platelet transfusion support; immune reconstitution studies done by flow cytometry.
Incidence of adverse events during phase II segment | Up to day +30 post HCT transplant
  Defined using the modified Bearman Scale and the National Cancer Institute Common Terminology Criteria for Adverse Events version 5.0 scale.
Acute GVHD biomarkers | Up to 2 years
JAK-regulated pro-inflammatory cytokines | Up to 2 years
STAT3 phosphorylation | Up to 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Haris Ali, Principal Investigator — City of Hope Medical Center
Locations (1):
- City of Hope Medical Center, Duarte, California, United States